CLINICAL TRIAL: NCT03403205
Title: A Phase 3, Randomized, Rater-Blinded, Multi-Center Study to Evaluate the Efficacy and Safety of ALXN1840 Administered for 48 Weeks Versus Standard of Care in Patients With Wilson Disease Aged 12 Years and Older, With an Extension Period of up to 60 Months
Brief Title: Efficacy and Safety of ALXN1840 Administered for 48 Weeks Versus Standard of Care in Participants With Wilson Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to terminate the program
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WTX101-301; 2017-004135-36 (EudraCT Number)
Record Dates: First submitted 2017-12-19; First posted 2018-01-18 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Wilson Disease
Keywords: Wilson Disease; ALXN1840; Copper
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — tetrathiomolybdate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study is rater-blinded for the Unified Wilson Disease Rating Scale (UWDRS) assessment only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALXN1840 (Experimental): ALXN1840 was administered orally for 48 weeks at doses ranging from 15 milligrams (mg) every other day (QOD) up to a titrated dose of 60 mg daily.
  Participants who completed the Primary Evaluation Period had the option to participate in the up to 60-month Extension Period.
  Interventions: Drug: ALXN1840
- Standard of Care (SoC) Medication (Active Comparator): SoC medication was administered for 48 weeks. Participants who completed the Primary Evaluation Period had the option to participate in the up to 60-month Extension Period.
  Interventions: Drug: SoC Therapy

INTERVENTIONS:
Drug: ALXN1840 — ALXN1840 administered orally in 15 mg tablets
  Other Names: Formerly named WTX101; Tiomolibdic acid; Tiomolibdate choline; Bis-choline tetrathiomolybdate
  Arms: ALXN1840
Drug: SoC Therapy — Depending on the site/region, participants randomized to receive SoC treatment will receive trientine, penicillamine, Zinc, or a combination of these medicines, administered according to standard regimens.
  Arms: Standard of Care (SoC) Medication

SUMMARY:
The study will evaluate the efficacy and safety of ALXN1840 (formerly called WTX101) administered for 48 weeks compared to standard of care (SoC) in Wilson Disease (WD) participants aged 12 and older in the Primary Evaluation Period. In addition, efficacy and safety will be evaluated during an optional 60-month Extension Period.

DETAILED DESCRIPTION:
The study consists of 2 cohorts. Cohort 1: Participants who have received SoC therapy for > 28 days and Cohort 2: Participants who are treatment-naïve or who have received SoC therapy for ≤ 28 days.

All enrolled participants were randomized by cohort in a 2:1 ratio to treatment with ALXN1840 or SoC (either as continued therapy in Cohort 1 or as continued or initial therapy in Cohort 2).

ELIGIBILITY:
Key Inclusion Criteria:

* Established diagnosis of WD by Leipzig-Score ≥ 4
* Female participants of childbearing potential, if heterosexually active, must be willing to follow protocol-specified guidance for highly effective contraception starting at least 6 weeks before the Day 1 visit and continuing through 28 days after the last dose of either ALXN1840 or SoC
* Male participants, if heterosexually active, must be willing to follow protocol-specified guidance for highly effective contraception beginning at Day 1 visit and continuing through 90 days after last dose of either ALXN1840 or SoC

Key Exclusion Criteria:

* Decompensated hepatic cirrhosis
* MELD score > 13
* Modified Nazer score > 7
* Clinically significant gastrointestinal bleed within past 3 months
* Alanine aminotransferase > 2 X upper limit of normal (ULN) for participants treated for > 28 days with WD therapy (Cohort 1)
* Alanine aminotransferase > 5 X ULN for treatment-naïve participants or participants who have been treated for ≤ 28 days (Cohort 2)
* Marked neurological disease requiring either nasogastric feeding or intensive inpatient medical care
* Hemoglobin < 9 grams/deciliter
* History of seizure activity within 6 months prior to informed consent
* Pregnant (or women who are planning to become pregnant) or breastfeeding women
* Active infection with hepatitis B virus (positive hepatitis B surface antigen) or C virus or seropositivity for human immunodeficiency virus (HIV)
* Previous treatment with tetrathiomolybdate
* Participants with end-stage renal disease on dialysis (chronic kidney disease stage 5) or creatinine clearance < 30 milliliter/minute

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene S. Swenson, M.D., Ph.D., Study Director — Alexion Pharmaceuticals, Inc.
Locations (51):
- United States (6):
  - Research Site, Los Angeles, California
  - Research Site, New Haven, Connecticut
  - Research Site, Chicago, Illinois
  - Research Site, Ann Arbor, Michigan
  - Research Site, Houston, Texas
  - Research Site, Seattle, Washington
- Australia (3):
  - Research Site, Adelaide
  - Research Site, Concord
  - Research Site, Parkville
- Austria (3):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Vienna
- Research Site, Toronto, Ontario, Canada
- Research Site, Prague, Czechia
- Research Site, Århus N, Denmark
- France (2):
  - Research Site, Bron
  - Research Site, Paris
- Germany (3):
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Leipzig
- Research Site, Hong Kong, Hong Kong
- Research Site, Budapest, Hungary
- Israel (2):
  - Research Site, Jerusalem
  - Research Site, Ramat Gan
- Japan (8):
  - Research Site, Chiba
  - Research Site, Kumamoto
  - Research Site, Kurume-shi
  - Research Site, Matsuyama
  - Research Site, Meguro-ku
  - Research Site, Sapporo
  - Research Site, Takatsuki-shi
  - Research Site, Yokohama
- Research Site, Grafton, New Zealand
- Research Site, Warsaw, Poland
- Russia (3):
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Saint Petersburg
- Research Site, Belgrade, Serbia
- Research Site, Singapore, Singapore
- Research Site, Daegu, South Korea
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Málaga
  - Research Site, Sabadell
- Taiwan (2):
  - Research Site, Taipei
  - Research Site, Taoyuan
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
- United Kingdom (3):
  - Research Site, Edgbaston
  - Research Site, Guildford
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=WTX101-301&attachmentIdentifier=7e63eb7b-ff32-4ef3-ba97-94d6dd3d86cd&fileName=wtx101-301-CSR_Synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of 2 periods: Primary Evaluation Period (PEP) and Open-label Extension (OLE) Period. Participants who completed the 48-week PEP were offered the opportunity to continue treatment in an up to 60-month Extension. A total of 214 participants were randomized; 207 participants were treated in the PEP.
Pre-assignment Details: Participants were randomized, stratified by cohort, in a 2:1 ratio to treatment with ALXN1840 or continued treatment with Standard of Care (SoC). Two cohorts were defined. Cohort 1: participants previously treated with SoC for >28 days; Cohort 2: participants who were treatment naïve or previously treated with SoC for ≤28 days. Participants who completed participation in Study WTX101-201 (NCT02273596) were offered the opportunity to participate in the Study WTX101-301 OLE Period.
Groups:
- Cohort 1: ALXN1840: Participants in Cohort 1 (who received SoC therapy, that is, chelation therapy with penicillamine or trientine, zinc therapy, or a combination of both chelation and zinc therapy for >28 days) received titrated doses of ALXN1840 orally for up to 48 weeks in PEP. Participants who completed the 48-week PEP were offered the opportunity to participate in the OLE Period and continued to receive ALXN1840 for up to 60 months.
- Cohort 1: SoC Therapy: Participants in Cohort 1 (who received SoC therapy, that is, chelation therapy with penicillamine or trientine, zinc therapy, or a combination of both chelation and zinc therapy for >28 days) continued to receive SoC therapy according to the local package label for up to 48 weeks in PEP. Participants who completed the 48-week PEP were offered the opportunity to participate in the OLE Period and received ALXN1840 for up to 60 months.
- Cohort 2: ALXN1840: Participants in Cohort 2 (who were treatment naïve or who received SoC therapy for ≤28 days) received titrated doses of ALXN1840 orally for up to 48 weeks in PEP. Participants who completed the 48-week PEP were offered the opportunity to participate in the OLE Period and continued to receive ALXN1840 for up to 60 months.
- Cohort 2: SoC Therapy: Participants in Cohort 2 (who were treatment naïve or who received SoC therapy for ≤28 days) received SoC therapy according to the local package label for up to 48 weeks in PEP. Participants who completed the 48-week PEP were offered the opportunity to participate in the OLE Period and received ALXN1840 for up to 60 months.
- Cohort 1: WTX101-201- ALXN1840; Cohort 2: WTX101-201- ALXN1840: Participants who received ALXN1840 during Study WTX101-201 (NCT02273596) continued to receive ALXN1840 for up to 60 months in the OLE period of this study.
Period: Primary Evaluation Period (48 Weeks)
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy | Cohort 1: WTX101-201- ALXN1840 | Cohort 2: WTX101-201- ALXN1840
Started | 105 | 56 | 37 | 16 | 0 | 0
Received at Least 1 Dose of Study Drug | 104 | 56 | 33 | 14 | 0 | 0
Completed PEP, Enter Extension | 89 | 49 | 28 | 12 | 0 | 0
Completed PEP, Not Into Extension | 4 | 3 | 1 | 1 | 0 | 0
Completed | 93 | 52 | 29 | 13 | 0 | 0
Not Completed | 12 | 4 | 8 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 2 | 1 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 1 | 0 | 4 | 2 | 0 | 0
Period: Extension Period (Up to 60 Months)
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy | Cohort 1: WTX101-201- ALXN1840 | Cohort 2: WTX101-201- ALXN1840
Started | 89 | 49 | 28 | 12 | 8 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 1
Not Completed | 89 | 49 | 28 | 12 | 8 | 10
Not completed — Withdrawal by Subject | 6 | 7 | 2 | 1 | 0 | 2
Not completed — Adverse Event | 6 | 3 | 1 | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 66 | 32 | 21 | 10 | 7 | 8
Not completed — Other than specified | 5 | 5 | 3 | 0 | 1 | 0
Not completed — Physician Decision | 2 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all randomized participants who received at least 1 dose of randomized treatment.
  The Extension Analysis Set included all participants who entered the Extension Period and received at least 1 dose of ALXN1840 in the Extension Period. This included the participants who rolled over from Study WTX101-201.
Groups:
- Cohort 1: ALXN1840: Participants in Cohort 1 (who received SoC therapy, that is, chelation therapy with penicillamine or trientine, zinc therapy, or a combination of both chelation and zinc therapy for >28 days) received titrated doses of ALXN1840 orally for up to 48 weeks.
- Cohort 1: SoC Therapy: Participants in Cohort 1 (who received SoC therapy, that is, chelation therapy with penicillamine or trientine, zinc therapy, or a combination of both chelation and zinc therapy for >28 days) continued to receive SoC therapy for up to 48 weeks according to the local package label.
- Cohort 2: ALXN1840: Participants in Cohort 2 (who were treatment naïve or who received SoC therapy for ≤28 days) received titrated doses of ALXN1840 orally for up to 48 weeks.
- Cohort 2: SoC Therapy: Participants in Cohort 2 (who were treatment naïve or who received SoC therapy for ≤28 days) received/continued to receive SoC therapy for up to 48 weeks according to the local package label.
- Cohort 1: WTX101-201- ALXN1840; Cohort 2: WTX101-201- ALXN1840: Participants who received ALXN1840 during Study WTX101-201 (NCT02273596) continued to receive ALXN1840 for up to 60 months.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy | Cohort 1: WTX101-201- ALXN1840 | Cohort 2: WTX101-201- ALXN1840 | Total
Number analyzed (Participants) | 104 | 56 | 33 | 14 | 8 | 11 | 226
Age, Customized [Count of Participants; unit: Participants]
  ≥12 years - <18 years | 10 | 4 | 2 | 2 | 0 | 0 | 18
  ≥18 years - <65 years | 92 | 50 | 31 | 12 | 7 | 11 | 203
  ≥65 years | 2 | 2 | 0 | 0 | 1 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 30 | 9 | 3 | 3 | 7 | 98
  Male | 58 | 26 | 24 | 11 | 5 | 4 | 128
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 19 | 13 | 5 | 0 | 1 | 1 | 39
  Race: Black or African American | 1 | 2 | 0 | 0 | 0 | 0 | 3
  Race: White | 80 | 41 | 27 | 12 | 7 | 9 | 176
  Race: Other | 3 | 0 | 0 | 2 | 0 | 0 | 5
  Race: Unknown | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Race: Not Reported | 1 | 0 | 0 | 0 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 2 | 1 | 0 | 7
  Not Hispanic or Latino | 101 | 54 | 32 | 11 | 7 | 11 | 216
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Daily Mean Area Under The Effect-time Curve (AUEC) of Directly Measured Non-ceruloplasmin-bound Copper (dNCC) From 0 to 48 Weeks (dNCC AUEC0-48W)
Description: dNCC is the directly quantified copper not bound to ceruloplasmin, obtained by inductively coupled plasma mass spectrometry after immunocapture and removal of ceruloplasmin. Baseline was defined as last non-missing value on or before first study drug administration. Least square (LS) mean and standard error (SE) was calculated using analysis of covariance (ANCOVA).
Time Frame: Baseline to Week 48
Population: Full analysis set included all randomized participants who received at least 1 dose of randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: micromoles (µmol)*hours (hr)/liter (L)
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 104 | 56 | 33 | 14
micromoles (µmol)*hours (hr)/liter (L) | 2.50 (0.150) [lower limit 0.150] | 0.87 (0.204) [lower limit 0.204] | 4.76 (0.319) [lower limit 0.319] | 0.96 (0.487) [lower limit 0.487]
Statistical Analysis 1: Comparison: Cohort 1: ALXN1840 vs Cohort 1: SoC Therapy; Analysis was performed using ANCOVA model, which included treatment, cohort, and baseline value. Missing imputation was performed: 1) for intermediate missing, interpolation was used to fill out missing values. 2) For participants who die, baseline dNCC was carried forward from discontinuation to week 48. 3) For others, multiple imputation was used to impute missing dNCC assuming data were missing not at random; Test type: Other; p < 0.0001, ANCOVA — Test was performed at a significance level of 0.05; LS Mean Difference = 1.64, 95% CI 2-sided [1.14 to 2.13], Standard Error of Mean 0.254
Statistical Analysis 2: Comparison: Cohort 2: ALXN1840 vs Cohort 2: SoC Therapy; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, ANCOVA — Test was performed at a significance level of 0.05; LS Mean Difference = 3.79, 95% CI 2-sided [2.65 to 4.94], Standard Error of Mean 0.584

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant administered the study drug and which did not necessarily have a causal relationship with this treatment. TEAEs were defined as those AEs with onset after the first dose of randomized treatment or existing events that worsened in severity after the first dose of randomized treatment. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to Week 48
Population: Safety analysis set included all participants who received at least 1 dose of randomized treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 104 | 56 | 33 | 14
Participants | 89 | 41 | 30 | 12

3. Secondary Outcome: Change From Baseline in the Unified Wilson Disease Rating Scale (UWDRS) Part II Total Score at Week 48
Description: The UWDRS comprises 3 parts: UWDRS Part I (level of consciousness, item 1), UWDRS Part II (a patient-reported review of daily activity items [disability], items 2 to 11 [10 items in total]), and UWDRS Part III (a detailed neurological examination, items 12 to 34 [23 items in total]). The UWDRS Part II total score was calculated as the sum of Question 2 to Question 11 (each question has range 0 [none] to 4 [severe]). The UWDRS Part II total score ranges from 0 (no disability) to 40 (severe disability), with lower score indicating improvement in condition and a better outcome. Change from baseline was calculated as: postbaseline assessment value - baseline assessment value when both values were not missing.
Time Frame: Baseline, Week 48
Population: Full analysis set included all randomized participants who received at least 1 dose of randomized treatment. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 92 | 50 | 29 | 12
units on a scale | -0.7 (2.75) [lower limit 2.75] | 0.0 (2.31) [lower limit 2.31] | -0.5 (3.23) [lower limit 3.23] | -1.8 (4.63) [lower limit 4.63]

4. Secondary Outcome: Change From Baseline in UWDRS Part III Total Score at Week 48
Description: The UWDRS comprises 3 parts: UWDRS Part I (level of consciousness, item 1), UWDRS Part II (a patient-reported review of daily activity items [disability], items 2 to 11 [10 items in total]), and UWDRS Part III (a detailed neurological examination, items 12 to 34 [23 items in total]). The UWDRS Part I and III was assessed by a neurologist who was blinded to the treatment randomization. The UWDRS Part III total score was calculated as the sum of Question 12 to Question 34. The UWDRS Part III total score ranges from 0 (normal) to 175 (severe disease), with lower score indicating improvement in condition and a better outcome. Change from baseline was calculated as: postbaseline assessment value - baseline assessment value when both values were not missing.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 91 | 49 | 28 | 11
units on a scale | -2.24 (7.458) [lower limit 7.458] | -1.59 (6.188) [lower limit 6.188] | -2.06 (9.843) [lower limit 9.843] | 1.55 (5.889) [lower limit 5.889]

5. Secondary Outcome: Change From Baseline in UWDRS Part III Functional Subscale Score at Week 48
Description: UWDRS Part III Functional Subscale consists of speech, handwriting, arising from chair, and gait from UWDRS Part III. The standardized score of the first 3 items ranges from 0 (normal) to 10 (worst), and standardized transformed score of gait ranges from 0 (normal) to 10 (worst). The average of these scores was used to create the Part III Functional Subscale with a range of 0 (normal) - 10 (worst) with higher scores indicating more functional disability.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 91 | 49 | 28 | 11
units on a scale | -0.165 (0.7620) [lower limit 0.7620] | -0.102 (0.5467) [lower limit 0.5467] | -0.090 (0.8464) [lower limit 0.8464] | 0.227 (0.4214) [lower limit 0.4214]

6. Secondary Outcome: Change From Baseline in UWDRS Part III Individual Items/Subscales (Speech, Handwriting, Arising From a Chair, and Gait) Score at Week 48
Description: UWDRS Part III individual items speech, handwriting, arising from chair, and gait are reported here. For speech (Question 12), original score ranges from 0 (normal) to 4 (unintelligible). For handwriting (Question 20), original score ranges from 0 (normal) to 4 (cannot hold a pen). For arising from chair (Question 27), original score ranges from 0 (normal) to 4 (unable to arise without help). For gait (Question 29), the original score (range: 0 [normal] to 10 [severe condition]) was calculated by summing subscores (0 [normal] to 4 [severe]) of Part A (Right and Left Leg dystonia), B (Ataxia), and C (Parkinsonism).
Time Frame: Baseline, Week 48
Population: Full analysis set included all randomized participants who received at least 1 dose of randomized treatment. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 91 | 49 | 28 | 11
units on a scale
  Speech | -0.1 (0.50) | 0.0 (0.35) | -0.1 (0.52) | 0.1 (0.54)
  Handwriting: number analyzed (Participants) | 91 | 48 | 28 | 11
  Handwriting | -0.2 (0.63) | -0.1 (0.48) | 0.1 (0.60) | 0.2 (0.40)
  Arising from a chair | 0.0 (0.45) | -0.1 (0.56) | 0.0 (0.27) | 0.0 (0.00)
  Gait | -0.03 (1.317) | 0.00 (1.141) | -0.18 (0.945) | 0.23 (0.754)

7. Secondary Outcome: Clinical Global Impression-Improvement Scale (CGI-I) Score at Week 48
Description: The CGI-I is a 7-point scale where the clinician assessed how much participant's illness improved or worsened relative to a Baseline state at the beginning of the intervention and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 92 | 50 | 27 | 12
units on a scale | 3.4 (0.89) [lower limit 0.89] | 3.8 (0.80) [lower limit 0.80] | 3.1 (1.06) [lower limit 1.06] | 3.2 (1.34) [lower limit 1.34]

8. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity Scale (CGI-S) Score at Week 48
Description: The CGI-S is a 7-point scale where the investigator rated severity of participant's illness at the time of assessment, relative to the investigator's past experience with participants who have the same diagnosis. Considering total clinical experience, a participant was assessed on severity of illness at time of rating as: 1, normal, not at all ill; 2, borderline ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 89 | 47 | 27 | 11
units on a scale | -0.4 (0.79) [lower limit 0.79] | -0.1 (0.73) [lower limit 0.73] | -0.6 (1.11) [lower limit 1.11] | -0.5 (1.21) [lower limit 1.21]

9. Secondary Outcome: Change From Baseline in Model for End-Stage Liver Disease (MELD) Score at Week 48
Description: The MELD score uses the participant's values for bilirubin, creatinine, and the international normalized ratio (INR). The initial MELD score (MELD[i]) is calculated according to the following formula: MELD(i) = 3.78*ln[serum bilirubin (mg/dL)] + 11.2*ln[INR] + 9.57*ln[serum creatinine (mg/dL)] + 6.43. Creatinine, bilirubin, and INR values less than 1.0 are set to 1.0 and creatinine values greater than 4.0 are set to 4.0 when calculating MELD(i). Additionally, creatinine, bilirubin, and INR are rounded to the 10th decimal place prior to performing the calculation. The initial MELD score is then rounded to the nearest integer. The MELD score ranges from 6 (least sick) - 40 (most sick), with higher values indicating more advanced disease.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 86 | 49 | 28 | 11
units on a scale | -0.1 (1.85) [lower limit 1.85] | 0.1 (1.32) [lower limit 1.32] | -0.7 (1.61) [lower limit 1.61] | 0.2 (1.25) [lower limit 1.25]

10. Secondary Outcome: Absolute Change From Baseline in Calculated Non-Ceruloplasmin Bound Copper (cNCC) or Calculated Non-Ceruloplasmin Bound Copper Corrected (cNCCcorrected) in Plasma at Week 48
Description: cNCC = Plasma Total Copper (Cu) [micrograms (µg)/L]-(3.15*ceruloplasmin [milligrams (mg)/L])/63.5 [µg/µmol] For ALXN1840-treated participants, cNCC in plasma corrected for amount of Cu bound to ALXN1840 tripartite complex (TPC) cNCCcorrected = (√cNCC- 0.993)2√Mo, (Mo= molybdenum). In calculation of cNCC and cNCCcorrected following rules apply: - For plasma total Cu concentration <lower limit of quantification (LLOQ), cNCC was considered missing (LLOQ = 20 nanograms [ng]/mL); - Serum ceruloplasmin concentration values <LLOQ are set to 0 (LLOQ = 22.5 mg/L); - Plasma total Mo concentration values <LLOQ are set to 0 (LLOQ = 1 ng/L); - If cNCC calculation produces a negative result, cNCC was considered missing and cNCCcorrected was not derived; - cNCCcorrected was set to 0 when 0.993√Mo > √cNCC.
Time Frame: Baseline, Week 48
Population: Full analysis set: all randomized participants who received at least 1 dose of study drug. 'Overall number of participants analyzed'= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 63 | 29 | 26 | 10
µmol/L | -0.72 (1.107) [lower limit 1.107] | 0.64 (2.769) [lower limit 2.769] | -1.95 (1.536) [lower limit 1.536] | -1.51 (2.361) [lower limit 2.361]

11. Secondary Outcome: Percent Change From Baseline in cNCC or cNCCcorrected in Plasma at Week 48
Description: cNCC [µmol/L] = Plasma Total Cu [µg/L]-(3.15*ceruloplasmin [mg/L])/63.5 [µg/µmol] For ALXN1840-treated participants, cNCC in plasma was corrected for amount of Cu bound to the ALXN1840 TPC using square root-based cNCC correction method: cNCCcorrected = (√cNCC- 0.993)2√Mo, where Mo = molybdenum. In calculation of cNCC and cNCCcorrected following rules apply: - For plasma total Cu concentration values <LLOQ, cNCC was considered missing (LLOQ = 20 ng/mL); - Serum ceruloplasmin concentration values <LLOQ are set to 0 (LLOQ = 22.5 mg/L); - Plasma total Mo concentration values <LLOQ are set to 0 (LLOQ = 1 ng/L); - In cases where cNCC calculation produces a negative result, cNCC was considered missing and cNCCcorrected was not derived; - cNCCcorrected was set to 0 when 0.993√Mo > √cNCC.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 60 | 28 | 26 | 10
percent change | -7.7 (263.20) [lower limit 263.20] | 104.6 (292.11) [lower limit 292.11] | -64.0 (42.88) [lower limit 42.88] | -44.3 (68.82) [lower limit 68.82]

12. Secondary Outcome: cNCC/cNCCcorrected Responder at Week 48
Description: cNCC/cNCCcorrected responder was defined as participants who achieved or maintained normalized cNCC/cNCCcorrected concentration (0.8-2.3 μmol) within (at or before) 48 weeks or reached a reduction of at least 25% in cNCC/cNCCcorrected within 48 weeks. Thus, a participant was considered a cNCC/cNCCcorrected responder if they met at least 1 of the following criteria: - Achieved normalized cNCC/cNCCcorrected concentration for 2 consecutive measurements within 48 weeks, for participants who had elevated cNCC concentrations at baseline; - Maintained normalized cNCC/cNCCcorrected concentration within 48 weeks, for participants who had normal cNCC concentrations at baseline; - Reached a reduction of at least 25% in cNCC/cNCCcorrected for 2 consecutive measurements within 48 weeks.
Time Frame: Week 48
Population: Full analysis set included all randomized participants who received at least 1 dose of randomized treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ALXN1840 | Cohort 1: SoC Therapy | Cohort 2: ALXN1840 | Cohort 2: SoC Therapy
Number analyzed (Participants) | 104 | 56 | 33 | 14
Participants | 101 | 39 | 33 | 13

ADVERSE EVENTS:
Time Frame: For PEP participants: From Primary Evaluation Period Baseline up to Primary Evaluation Period Week 48/Early Termination; For OLE and WTX101-201 participants: From Extension Period Week 1 up to Extension Period Week 268/Early Termination
Description: Safety analysis set included all participants who received at least 1 dose of randomized treatment.
Groups:
- PEP Cohort 1: ALXN1840: Participants in Cohort 1 (who received SoC therapy, that is, chelation therapy with penicillamine or trientine, zinc therapy, or a combination of both chelation and zinc therapy for >28 days) received titrated doses of ALXN1840 orally for up to 48 weeks.
- PEP Cohort 1: SoC Therapy: Participants in Cohort 1 (who received SoC therapy, that is, chelation therapy with penicillamine or trientine, zinc therapy, or a combination of both chelation and zinc therapy for >28 days) continued to receive SoC therapy for up to 48 weeks according to the local package label.
- PEP Cohort 2: ALXN1840: Participants in Cohort 2 (who were treatment naïve or who received SoC therapy for ≤28 days) received titrated doses of ALXN1840 orally for up to 48 weeks.
- PEP Cohort 2: SoC Therapy: Participants in Cohort 2 (who were treatment naïve or who received SoC therapy for ≤28 days) received SoC therapy for up to 48 weeks according to the local package label.
- OLE Cohort 1: ALXN1840: Participants in Cohort 1 (who received SoC therapy, that is, chelation therapy with penicillamine or trientine, zinc therapy, or a combination of both chelation and zinc therapy for >28 days) who completed the 48-week PEP of study WTX101-301 were offered the opportunity to participate in the OLE Period and continued to receive ALXN1840 for up to 60 months.
- OLE Cohort 1: SoC Therapy: Participants in Cohort 1 (who received SoC therapy, that is, chelation therapy with penicillamine or trientine, zinc therapy, or a combination of both chelation and zinc therapy for >28 days) who completed the 48-week PEP of study WTX101-301 were offered the opportunity to participate in the OLE Period and received ALXN1840 for up to 60 months.
- OLE Cohort 2: ALXN1840: Participants in Cohort 2 (who were treatment naïve or who received SoC therapy for ≤28 days) who completed the 48-week PEP were offered the opportunity to participate in the OLE Period and continued to receive ALXN1840 for up to 60 months.
- OLE Cohort 2: SoC Therapy: Participants in Cohort 2 (who were treatment naïve or who received SoC therapy for ≤28 days) who completed the 48-week PEP were offered the opportunity to participate in the OLE Period and received ALXN1840 for up to 60 months.
Arm/Group | PEP Cohort 1: ALXN1840 | PEP Cohort 1: SoC Therapy | PEP Cohort 2: ALXN1840 | PEP Cohort 2: SoC Therapy | OLE Cohort 1: ALXN1840 | OLE Cohort 1: SoC Therapy | OLE Cohort 2: ALXN1840 | OLE Cohort 2: SoC Therapy | Cohort 1: WTX101-201- ALXN1840 | Cohort 2: WTX101-201- ALXN1840
All-Cause Mortality (participants affected / at risk) | 1/104 | 0/56 | 1/33 | 0/14 | 1/89 | 0/49 | 0/28 | 0/12 | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 14/104 | 6/56 | 4/33 | 0/14 | 20/89 | 10/49 | 6/28 | 3/12 | 2/8 | 3/11
Other Adverse Events (participants affected / at risk) | 46/104 | 18/56 | 16/33 | 7/14 | 45/89 | 32/49 | 10/28 | 4/12 | 6/8 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEP Cohort 1: ALXN1840 (N=104) | PEP Cohort 1: SoC Therapy (N=56) | PEP Cohort 2: ALXN1840 (N=33) | PEP Cohort 2: SoC Therapy (N=14) | OLE Cohort 1: ALXN1840 (N=89) | OLE Cohort 1: SoC Therapy (N=49) | OLE Cohort 2: ALXN1840 (N=28) | OLE Cohort 2: SoC Therapy (N=12) | Cohort 1: WTX101-201- ALXN1840 (N=8) | Cohort 2: WTX101-201- ALXN1840 (N=11)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepato-lenticular degeneration (Congenital, familial and genetic disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurological decompensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unevaluable event (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex hepatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sports injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurological symptom (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEP Cohort 1: ALXN1840 (N=104) | PEP Cohort 1: SoC Therapy (N=56) | PEP Cohort 2: ALXN1840 (N=33) | PEP Cohort 2: SoC Therapy (N=14) | OLE Cohort 1: ALXN1840 (N=89) | OLE Cohort 1: SoC Therapy (N=49) | OLE Cohort 2: ALXN1840 (N=28) | OLE Cohort 2: SoC Therapy (N=12) | Cohort 1: WTX101-201- ALXN1840 (N=8) | Cohort 2: WTX101-201- ALXN1840 (N=11)
Nausea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 2 (2) | 2 (2) | 6 (10) | 3 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (14) | 10 (12) | 4 (4) | 2 (2) | 9 (14) | 6 (6) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 19 (24) | 1 (1) | 1 (1) | 1 (1) | 8 (13) | 13 (16) | 2 (5) | 1 (1) | 1 (8) | 1 (1)
Headache (Nervous system disorders) | 7 (7) | 3 (8) | 4 (5) | 3 (3) | 8 (10) | 6 (13) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 6 (8) | 1 (3) | 4 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 9 (12) | 2 (2) | 4 (4) | 1 (1) | 4 (5) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 22 (23) | 12 (12) | 6 (7) | 4 (5) | 2 (2) | 7 (7)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (13) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT03403205/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT03403205/SAP_001.pdf